CLINICAL TRIAL: NCT05282485
Title: Mitigating Infectious Morbidity and Growth Deficits in HIV Exposed Uninfected infanTs With Human Milk Oligosaccharides
Acronym: MIGH-T MO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: University of Stellenbosch (Other); University of California, Los Angeles (Other); University of California, San Diego (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Rupak Shivakoti, Assistant Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AAAT8393; R01HD105492 (NIH)
Record Dates: First submitted 2022-02-10; First posted 2022-03-16 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: HIV; Infant Morbidity; Breast Feeding
Keywords: HIV; Infant Morbidity; Infant Growth; Breastmilk; Probiotic; Synbiotic; HIV-exposed Uninfected Infants; B. infantis; Human Milk Oligosaccharides; 2'-Fucosyllactose; Infant neurodevelopment
MeSH Terms: conditions — Breast Feeding | interventions — Synbiotics; maltodextrin

STUDY DESIGN:
Intervention Model Description: This study will recruit 144 women living with HIV and their HIV-exposed uninfected children (72 will receive the interventional product and 72 will receive the placebo). All of the women in the study will have breastfed or are currently breastfeeding their children.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotic Group (Experimental): A synbiotic combining 2'-Fucosyllactose (2'-FL) human milk oligosaccharides (HMO) with B.infantis (probiotic) will be administered to infants from 4 to 24 weeks of age.
  Interventions: Dietary Supplement: Synbiotic
- Placebo Group (Placebo Comparator): Maltodextrin will be administered to infants from 4 to 24 weeks of age.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Synbiotic — Synbiotic (2'-FL HMO + B. infantis probiotics)
  Arms: Synbiotic Group
Dietary Supplement: Maltodextrin — Maltodextrin
  Arms: Placebo Group

SUMMARY:
Primary Objective:

* To evaluate the effects of synbiotics on infectious morbidity and growth while it is in place from 4 to 24 weeks of age.
* To evaluate the effects of synbiotics on infectious morbidity and growth from 4 to 48 weeks of age.

Secondary Objectives:

* To evaluate the effects of synbiotics on growth from 4 to 72 weeks of age.
* To evaluate the effects of synbiotics on infant neurodevelopment at 48 and 72 weeks of age.
* To evaluate the effects of synbiotics on biological measurements while it is in place from 4 to 24 weeks of age.
* To evaluate the effects of synbiotics on biological measurements from 4 to 48 weeks of age.
* To evaluate the effects of synbiotics on gut microbiome and fecal short chain fatty acids from 4 to 72 weeks of age.
* To investigate feasibility, acceptance, tolerability, and behavioral adherence with the intervention.
* To investigate whether the synbiotics reduces infectious morbidity and improves growth in CHEU relative to CHUU.
* To investigate whether infant gut microbiota composition, maturity and function, and markers of inflammation and HMOs at baseline and over time are associated with morbidity and poor growth in CHEU and CHUU.

DETAILED DESCRIPTION:
Children who are HIV-exposed uninfected (CHEU), i.e., children born to mothers with HIV but who do not acquire HIV infection, have a higher risk of mortality, infectious morbidity, and growth deficits than children who are HIV-unexposed uninfected (CHUU), i.e., children whose mothers do not have HIV. Prior research has focused on breastfeeding and has pointed to changes in human milk oligosaccharides (HMOs) associated with maternal HIV infection that appear to influence the infant microbiome and thereby lead to these adverse outcomes. A randomized trial of an intervention which combines HMOs and probiotics in breastfed CHEU will be conducted in South Africa to evaluate whether this intervention has the potential to reduce excess infectious morbidity and growth faltering risks observed in CHEU. CHEU will be randomized 1:1 to either a) intervention (synbiotic: 2'-FL HMO + B. infantis probiotic) or b) placebo (Maltodextrin). The study intervention or placebo will be given from 4-24 weeks of age (total 20 weeks), followed by another 48 weeks of observation off study treatment. Both arms will be followed to 72 weeks of age for assessment of infant outcomes.

ELIGIBILITY:
Inclusion Criteria for Mothers:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Greater than 18 years of age
* For HIV-exposed uninfected children (CHEU): Mothers living with HIV documented based on medical record and with viral suppression (i.e., <400 copies/mL viral load) documented at delivery
* For HIV-unexposed uninfected children (CHUU): Mothers without HIV (document HIV-negative test result at delivery or screening)
* Women who initiated breastfeeding of their infant including:

  * Women who currently exclusively breastfeed their infants, or
  * Women who breastfed their infants for a period but are no longer breastfeeding, or
  * Women who are currently breastfeeding their infants in addition to feeding them formula milk or solids
* For women with HIV: Those currently on first-line standard of care antiretroviral therapy that was initiated a minimum of 12 weeks prior to delivery of the infant included in this study
* Participant has a cell phone that can be used for calls and messages
* Agreement to adhere to Lifestyle Considerations throughout study duration

Inclusion Criteria for Children:

* 3-6 weeks of age
* Delivered from a singleton pregnancy
* For children of mothers with HIV: At least one HIV diagnostic nucleic acid amplification test prior to enrollment which is negative and no positive test
* Child is well enough to have established full breastfeeding by the time of enrollment

Exclusion Criteria:

* Severe maternal or infant illness (e.g., maternal: tuberculosis, major psychiatric or neurological conditions; infant: any congenitally-acquired infections, major congenital anomalies)
* Use of immunomodulatory or immunosuppressive drugs in either mother or child prior to enrollment in the study
* For mothers with HIV: Mothers who are not currently receiving antiretroviral therapy or who are on regimens other than the currently recommended first-line standard of care in South Africa i.e., first-line dolutegravir- or efavirenz-based regimens.
* Children infected with HIV
* Mother or infant currently taking probiotics, prebiotics, or fiber supplements; or on any nutritional supplements (e.g., FM85) that impact the outcomes of interest
* Mother or infant currently taking antibiotics for more than 14 days, excluding preventative therapies
* Known allergic reactions to components of the treatment or placebo
* Any condition that, in the opinion of the study staff, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the aims of the study.

Ages: 3 Weeks to 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of infants with infectious morbidity from 4-24 weeks | 4-24 weeks of age
  Infectious morbidity data related to infectious respiratory or gastrointestinal morbidity will be compared between the two arms
Infant length for age Z scores (LAZ) from 4-24 weeks | 4-24 weeks of age
  Infant anthropometry will be recorded at each visit to calculate infant length for age Z scores (LAZ) will be compared between the two arms
Proportion of infants with infectious morbidity from 4-48 weeks | 4-48 weeks of age
  Infectious morbidity data related to infectious respiratory or gastrointestinal morbidity will be compared between the two arms
Infant length for age Z scores (LAZ) from 4-48 weeks | 4-48 weeks of age
  Infant anthropometry will be recorded at each visit to calculate infant length for age Z scores (LAZ) will be compared between the two arms

SECONDARY OUTCOMES:
Infant weight for age (WAZ) and weight for length (WLZ) Z scores from 4-24 weeks | 4-24 weeks of age
  Infant anthropometry will be recorded at each visit to calculate infant weight for age (WAZ) and weight for length (WLZ) Z scores and will be compared between the two arms
Infant weight for age (WAZ) and weight for length (WLZ) Z scores from 4-48 weeks | 4-48 weeks of age
  Infant anthropometry will be recorded at each visit to calculate infant weight for age (WAZ) and weight for length (WLZ) Z scores and will be compared between the two arms
Infant length for age (LAZ), weight for age (WAZ) and weight for length (WLZ) Z scores from 4-72 weeks | 4-72 weeks of age
  Infant anthropometry will be recorded at each visit to calculate infant length for age (LAZ), weight for age (WAZ) and weight for length (WLZ) Z scores and will be compared between the two arms
Infant microbiota-for-age Z scores (MAZ) | 4-72 weeks of age
  Infant microbiota-for-age Z scores (MAZ), a measure of infant microbiome maturity, will be compared between the two arms
Infant microbiota diversity | 4-72 weeks of age
  Microbiota diversity of taxa will be compared between the two arms
Infant microbiota relative abundance | 4-72 weeks of age
  Microbiota relative abundance of taxa will be compared between the two arms
Infant fecal short-chain fatty acid levels | 4-72 weeks of age
  Short-chain fatty acid (SCFA) levels in stool samples from infants will be compared between the two arms
Infant plasma metabolite levels | 4-24 weeks of age
  Unbiased metabolomics will be used to investigate whether metabolite levels and major metabolic pathways are different between the two arms
Infant plasma inflammatory markers and growth hormone levels | 4-48 weeks of age
  Levels of protein inflammatory markers and growth hormones will be measured using immunoassays and will be compared between the two arms
Infant plasma HMO levels | 4-24 weeks of age
  Infant HMO levels will be measured and compared between the two arms
Proportion of infants with Adverse Events (AEs)/Serious Adverse Event (SAEs) | Through 24 weeks of age
  Proportion of AE/SAEs will be recorded and compared between the two arms to assess the safety of the intervention
Proportion of infants with tolerability symptoms | Through 8 weeks of age
  Digestive tolerability will be assessed and compared between the two arms to assess the safety of the intervention
Proportion of infants with severe infectious morbidity | 4-48 weeks of age
  Severe infectious morbidity (i.e., those requiring hospitalizations) data related to infectious respiratory or gastrointestinal morbidity will be compared between the two arms
Infant neurodevelopment milestones | 48-72 weeks
  A comprehensive neurodevelopment assessment, i.e., Griffiths III scale, will be conducted on infants at weeks 48 and 72 and the proportion passing each milestone will be compared between the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Rupak Shivakoti, PhD, Principal Investigator — Columbia University Assistant Professor
Locations (1):
- Worcester Campus of Stellenbosch University (SU), Stellenbosch, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shivakoti R, Laughton B, Shafiq M, Schoeman E, Glashoff RH, Barnabas S, Fry S, Leu CS, Wang S, Bode L, Aldrovandi G, Kuhn L, Slogrove AL. Feasibility Study of a Powder-Based Supplement Intervention for a future Synbiotic Trial in Breastfed Children from South Africa. Res Sq [Preprint]. 2023 May 15:rs.3.rs-2842773. doi: 10.21203/rs.3.rs-2842773/v1. PMID 37293067
- [Derived] Shivakoti R, Slogrove AL, Laughton B, Shafiq M, Schoeman E, Glashoff RH, Leu CS, Wang S, Bode L, Aldrovandi G, Kuhn L. Mitigating Infectious morbidity and Growth deficits in HIV-exposed uninfected infanTs with human Milk Oligosaccharide (MIGH-T MO): a randomised trial protocol. BMJ Open. 2022 Dec 30;12(12):e069116. doi: 10.1136/bmjopen-2022-069116. PMID 36585139